CLINICAL TRIAL: NCT00014170
Title: Phase II Study Of ZD1839 (NSC 715055) In Newly Diagnosed Patients With Glioblastoma (Grade 4 Astrocytoma)
Brief Title: Gefitinib in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01855; N0074; CDR0000068511; NCCTG-N0074; U10CA025224 (NIH)
Record Dates: First submitted 2001-04-10; First posted 2003-06-10 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-06

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Gefitinib

ARMS (1):
- Treatment (gefitinib) (Experimental): Patients receive oral gefitinib daily. Courses repeat every 8 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gefitinib; Other: pharmacological study; Other: laboratory biomarker analysis; Other: questionnaire administration; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: gefitinib — Given orally
  Other Names: Iressa; ZD 1839
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies
Other: questionnaire administration — Ancillary studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
Biological therapies such as gefitinib may interfere with the growth of the tumor cells and slow the growth of glioblastoma multiforme. Phase II trial to study the effectiveness of gefitinib in treating patients who have newly diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine treatment effectiveness of gefitinib, in terms of response rate, time to progression, survival at 52 weeks, progression-free survival at 6 months, and overall survival, in patients with newly diagnosed glioblastoma multiforme.

II. Determine the toxic effects of this drug in these patients. III. Assess fatigue, depression, excessive daytime somnolence, and quality of life in patients treated with this drug.

IV. Assess individual variation in responses, pharmacokinetic parameters, and/or biological correlates due to genetic differences in enzymes involved in transport, metabolism, and/or mechanism of action of this drug in these patients.

V. Determine if the type of epidermal growth factor receptor affects tumor response and outcome in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive oral gefitinib daily. Courses repeat every 8 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, before each treatment course, every 4 months for 1 year, every 6 months for 4 years, and then annually for 5 years.

Patients are followed every 8 weeks until tumor progression and then every 3 months for 5 years and annually for up to 10 years. Patients removed from study treatment for reasons other than disease progression are followed every 4 months for 1 year, every 6 months for 4 years, and then annually for 5 years.

PROJECTED ACCRUAL: A total of 92 patients will be accrued for this study within 14 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed newly diagnosed WHO grade IV astrocytoma (glioblastoma multiforme) or gliosarcoma

  * No WHO grade III anaplastic astrocytoma, oligodendroglioma, or mixed oligoastrocytoma
* Completed standard external beam radiotherapy within the past 2-5 weeks

  * No evidence of tumor progression during radiotherapy
* Performance status - ECOG 0-2
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10.0 g/dL
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST no greater than 3 times ULN
* Creatinine no greater than 1.5 times ULN
* No other active malignancy
* No uncontrolled infection
* No other severe concurrent disease that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior chemotherapy (including polifeprosan 20 with carmustine implant) for this tumor
* See Disease Characteristics
* No prior stereotactic radiosurgery or interstitial brachytherapy
* No more than 15 weeks since prior surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2001-03; Primary Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Survival | 52 weeks
  The proportion of 'successes' will be estimated using the binomial point estimator (number of 'successes' divided by the total number of evaluable patients) and standard binomial 90% confidence interval estimates. In the unlikely event that accrual has not been completed before the interim analyses are performed, the Duffy-Santner lgorithm will be used to calculate 90% confidence intervals.

SECONDARY OUTCOMES:
Post-RT progression-time | From start of study therapy to date of disease progression or last follow-up, assessed up to 10 years
  Kaplan-Meier survival curves and logrank tests will be used.
Toxicity patterns assessed using NCI CTC version 2.0 | Up to 10 years
  Will be analyzed descriptively. Toxicity score calculated as the sum of the maximum toxicity grades recorded for each of the types of adverse reactions observed during the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Joon Uhm, Principal Investigator — North Central Cancer Treatment Group
Locations (1):
- North Central Cancer Treatment Group, Rochester, Minnesota, United States